CLINICAL TRIAL: NCT00388024
Title: A Pilot Feasibility Study of PET-CT Imaging in Patients With Cancer of the Head and Neck Treated With Definitive Chemoradiation
Brief Title: PET Scans and CT Scans in Patients With Locally Advanced Head and Neck Cancer Undergoing Chemotherapy and Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000504047; CCCWFU-60A05; CCCWFU-BG06-007
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma of Unknown Primary; Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the nasopharynx; stage III lymphoepithelioma of the oropharynx; squamous cell carcinoma of unknown primary; newly diagnosed carcinoma of unknown primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; untreated metastatic squamous neck cancer with occult primary; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the oropharynx
MeSH Terms: conditions — Neoplasms, Unknown Primary; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer patients about to be treated with radiation therapy: Patienta with histologically confirmed squamous cell or lymphoepithelioma of oral cavity, oropharynx, hypopharynx, larynx, nasopharynx, or unknown primary of the head and neck about to be treated with radiation therapy

SUMMARY:
RATIONALE: Imaging procedures, such as PET scan and CT scan, may help doctors predict a patient's response to treatment and plan the best treatment.

PURPOSE: This clinical trial is studying how well PET scans and CT scans show response to treatment in patients with locally advanced head and neck cancer undergoing chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of performing positron emission tomography-computed tomography (PET-CT) imaging for early discrimination of treatment response and post-therapy neck management in patients with locally advanced cancer of the head and neck treated with definitive chemoradiotherapy.

Secondary

* Perform semiquantitative analysis of tracer uptake in these patients using standard uptake values and qualitative analysis of tracer uptake using pure visual analysis.
* Determine the feasibility of distinguishing benign from malignant processes during initial tumor staging of these patients by whole-body PET-CT imaging.
* Correlate staging by whole-body PET-CT imaging with staging by standard CT/MRI, clinical exam, and pathologic specimen.
* Determine the feasibility of PET-CT imaging in these patients in treatment position for radiotherapy treatment planning, correlate the results with standard CT/MRI images, and record the differences.
* Perform PET-CT imaging in these patients during weeks 2 and 4 of chemoradiotherapy to evaluate the predictive value of response to treatment at these time points.
* Determine if the time interval for treatment monitoring at 6 and 12 weeks post chemoradiotherapy is important for the predictive value of PET-CT imaging.
* Evaluate patients with clinical or radiographic abnormalities worrisome for residual or recurrent disease with PET-CT imaging at 6 and 12 weeks post chemoradiotherapy to assess the need for additional therapies (i.e., neck dissection).

OUTLINE: This is a pilot study.

Patients receive fludeoxyglucose F 18 (FDG) IV over 90 seconds prior to the initial scan. Patients undergo whole-body computed tomography (CT) imaging with contrast followed by positron emission tomography (PET) imaging (approximately 1 hour after FDG injection) for initial staging and simulation for radiotherapy treatment planning. After PET-CT evaluation, patients with locoregional disease are recommended for standard-care chemoradiotherapy. Patients with evidence of M1 disease that is confirmed by CT/MRI and/or biopsy are treated at the discretion of the attending clinician. During chemoradiotherapy, patients undergo PET-CT imaging, as described above, at the beginning of week 2 and during week 4 for treatment monitoring and early detection of recurrent or residual disease. Follow-up PET-CT scans are performed, as described previously, at 6 weeks and then at 3 months after completion of chemoradiotherapy.

After completion of study procedures, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma or lymphoepithelioma of the head and neck, including any of the following sites:

  * Oral cavity
  * Oropharynx
  * Hypopharynx
  * Larynx
  * Nasopharynx
  * Unknown primary of the head and neck region
* Stage III or IV disease
* Definitive chemoradiotherapy with curative intent must be planned

PATIENT CHARACTERISTICS:

* Able to tolerate positron emission tomography (PET) imaging
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No poorly controlled diabetes mellitus (e.g., fasting glucose > 200 mg/dL) despite medication

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Prognostic value of positron emission tomography-computed tomography imaging in predicting clinical response at baseline, at weeks 2 and 4, and at week 6 post chemoradiotherapy | 3 months
  The results of the experimental scans will be compared to the response to radiation therapy as measured by routine scans at 6 weeks and 3 months after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Greven, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States